CLINICAL TRIAL: NCT04855201
Title: A Phase 1b Multiple Oral Dose Study to Evaluate the Pharmacological Effect, Safety and Tolerability of ASP0367 in Participants With Reduced Maximum Oxygen Uptake Due to Poor Systemic Oxygen Extraction
Brief Title: A Study to Evaluate ASP0367 in Participants With Reduced Maximum Oxygen Uptake Due to Poor Systemic Oxygen Extraction
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Lack of Pharmacological effect
Sponsor: Astellas Pharma Global Development, Inc. (Industry)
Responsible Party: Sponsor
Organization: Astellas Pharma Inc (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 0367-CL-1101
Record Dates: First submitted 2021-04-20; First posted 2021-04-22 (Actual); Last update posted 2025-04-16 (Actual); Status verified 2025-04

CONDITIONS: Reduced Maximum Oxygen Uptake Due to Poor Systemic Oxygen Extraction
Keywords: Maximum oxygen intake; Peak exercise; Bocidelpar

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Bocidelpar (ASP0367) (Experimental): Participants will receive Bocidelpar (ASP0367) once daily in the morning for 6 weeks.
  Interventions: Drug: Bocidelpar
- Placebo (Placebo Comparator): Participants will receive placebo once daily in the morning for 6 weeks.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Bocidelpar — Oral
  Other Names: MA-0211; ASP0367
  Arms: Bocidelpar (ASP0367)
Drug: Placebo — Oral
  Arms: Placebo

SUMMARY:
The purpose of this study is to to evaluate the effect of ASP0367 on improvement of aerobic capacity relative to placebo, as well as evaluate the safety and tolerability of ASP0367 relative to placebo. This study will also evaluate the effect of ASP0367 on improvement of other aerobic capacity parameters relative to placebo, as well as evaluate the effect of ASP0367 on improvement of functional capacity relative to placebo.

DETAILED DESCRIPTION:
The study will consist of a screening period (up to 27 days [approximately 4 weeks]), treatment period (up to 44 days [6 weeks]) and follow-up period (7 days [1 week]).

The study will be completed with an end-of-study visit (ESV). The ESV will take place 7 days (1 week) after the end-of-treatment on day 44 (week 6) or 7 days (1 week) after early discontinuation from the study.

The anticipated total duration of the study for each participant, including screening and follow-up, is approximately 75 days (11 week).

An interim analysis may be performed before the end of the study.

ELIGIBILITY:
Inclusion Criteria:

* Participant agrees and is able to adhere to the study requirements for the length of the study, including undergoing both aCPET and SHAPE Test.
* Participant has a body mass index (BMI) range of 17.0 to 36 kg/m^2, inclusive and weighs at least 50 kg (male participant) or 40 kg (female participant) at screening.
* Participants with reduced maximum oxygen uptake due to poor SOE, defined as peak exercise ([Ca-VO2])/[Hb]) ≤ 0.85 and VO2max < 85% predicted in the absence of a cardiac or pulmonary mechanical limit, determined by aCPET within 6 months prior to day 1 or participants with reduced maximum oxygen uptake due to poor SOE, defined as peak exercise ([Ca-VO2])/[Hb]) ≤ 0.85 and VO2max < 85% predicted in the absence of a cardiac or pulmonary mechanical limit, determined by historical aCPET within 45 months of screening and confirmed reduction in skeletal muscle citrate synthase activity.
* Female participant is not pregnant and at least 1 of the following conditions apply:

  * Not a woman of childbearing potential (WOCBP)
  * WOCBP who agrees to follow the contraceptive guidance from the time of informed consent through at least 28 days after final IP administration.
* Female participant must agree not to breastfeed starting at screening and throughout the study period and for 28 days after final IP administration.
* Female participant must not donate ova starting at first dose of IP and throughout the study period and for 28 days after final IP administration.
* Male participant with female partner(s) of childbearing potential (including breastfeeding partner[s]) must agree to use contraception throughout the treatment period and for 28 days after final IP administration.
* Male participant must not donate sperm during the treatment period and for 28 days after final IP administration.
* Male participant with pregnant partner(s) must agree to remain abstinent or use a condom for the duration of the pregnancy throughout the study period and for 28 days after final IP administration.
* Participant agrees not to participate in another interventional study while participating in the present study.

Exclusion Criteria:

* Participant has signs and/or symptoms due to a cerebellar, pyramidal, extrapyramidal or other nonmyopathic process (e.g., cerebellar dysfunctions, movement disorder) that would interfere in any nontrivial manner with aCPET or SHAPE Test.
* Participant has received any investigational therapy within 28 days or 5 half-lives, whichever is longer, prior to screening.
* Participant has any condition which makes the participant unsuitable for study participation.
* Participant has used moderate or strong inducers of CYP3A, CYP2C8 and CYP2C19 within the 3 months prior to day -1.
* Participant has cardiac troponin I (cTnI) > ULN (or cardiac troponin T > ULN if cTnI is not available) at screening.
* Participant has estimated glomerular filtration rate (eGFR) calculated by the modification of diet in renal disease equation < 60 mL/min per 1.73 m^2 at screening.
* Participant has at screening: total bilirubin (TBL) > upper limit of normal (ULN) or transaminase(s) (aspartate aminotransferase [AST] or alanine aminotransferase [ALT]) > ULN in the absence of elevations in creatine kinase.
* Participant has diabetes mellitus (types 1 or 2).
* Participant has mental conditions such as schizophrenia, bipolar disorder or major depressive disorder that has not been under control within 1 year prior to screening.
* Participant has severe behavioral or cognitive problems that preclude participation in the study.
* Participant has a history of suicide attempt, suicidal behavior or has any suicidal ideation within 1 year prior to screening that meets criteria at a level of 4 or 5 by using the Columbia-Suicide Severity Rating Scale (C-SSRS) or who is at significant risk to commit suicide.
* Participant has undergone an inpatient hospitalization within the 30 days prior to the randomization or has a planned hospitalization or a surgical procedure during the study, which may affect the study assessments.
* Participant has clinically significant respiratory disease (such as chronic obstructive pulmonary disease, cystic fibrosis, severe asthma, lung infections including tuberculosis, sarcoidosis, thoracic endometriosis, pulmonary fibrosis and lung cancers) and/or cardiac disease (medical history or current clinical findings) or prior interventional cardiac procedure (e.g., left heart catheterization which resulted in angioplasty/percutaneous coronary intervention, balloon valvuloplasty, etc.) within 3 months prior to randomization.
* Participant has a pacemaker, implantable cardioverter-defibrillator or cardiac resynchronization therapy device, or has a mean corrected QT interval using Fridericia's formula (QTcF) > 450 msec for male participants and > 470 msec for female participants at screening or randomization. If QTcF exceeds these limits, 1 additional triplicate ECG can be taken on the same day in order to determine the participant's eligibility.
* Participant has ECG evidence of acute ischemia, atrial fibrillation or active conduction system abnormalities at screening, with the exception of any of the following:

  * First degree atrioventricular (AV)-block
  * Second degree AV-block type 1 (Mobitz type 1/Wenckebach type)
  * Right bundle branch block
* Participant has a seizure disorder that may interfere with their ability to complete all study requirements.
* Participant has an active malignancy or any other cancer from which the participant has been disease-free for < 5 years.
* Participant has a solid organ transplant and is currently receiving treatment with therapy for immunosuppression.
* Participant has a positive serology test for human immunodeficiency virus, hepatitis B or hepatitis C infection at screening.
* Participant has previously received ASP0367.
* Participant has a history of active substance abuse within 1 year prior to randomization.
* Participant has smoked, used tobacco-containing products and nicotine or nicotine-containing products (e.g., electronic vapes) within 6 months prior to screening or the participant tests positive for cotinine at screening or on day -1.
* Participant has a history of consuming > 14 units for male participants or 7 units for female participants of alcoholic beverages per week within 6 months prior to screening or has a history of alcoholism or drug/chemical/substance abuse within 2 years prior to screening (note: 1 unit = 12 ounces of beer, 4 ounces of wine, 1 ounce of spirits/hard liquor) or the participant tests positive for alcohol at screening or on day -1.
* Participant has used any drugs of abuse, that are not prescribed for a medical diagnosis (amphetamines, barbiturates, benzodiazepines, cannabinoids, cocaine and/or opiates) within 3 months prior to day -1 or the participant tests positive for drugs of abuse without a prescription (amphetamines, barbiturates, benzodiazepines, cannabinoids, cocaine and/or opiates) at screening or on day -1.
* Participant has used any PPAR ligands such as fibrates and thiazolidinediones (e.g., clinofibrate, clofibrate, fenofibrate, gemfibrozil, pioglitazone, rosiglitazone) within 4 weeks prior to randomization.
* Participant has used mestinon within 2 weeks prior to randomization.
* Participant has initiated the use of coenzyme Q10 (CoQ10), carnitine, creatine or other mitochondrial-focused supplements within 4 weeks prior to randomization.
* Participant has initiated an exercise regimen within 4 weeks prior to randomization.
* Participant has a known or suspected hypersensitivity to ASP0367 or any components of the formulation used.
* Participant has a positive result for SARS-CoV-2 polymerase chain reaction (PCR) test at screening.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 31 (Actual)
Dates: Start 2021-06-14 (Actual); Primary Completion 2022-12-16 (Actual); Study Completion 2022-12-16 (Actual)

PRIMARY OUTCOMES:
Change from baseline in maximum oxygen uptake at peak exercise (VO2max) during Advanced Cardiopulmonary Exercise Test (aCPET) | Baseline and Week 6
  V02max is defined as maximum amount of oxygen body can utilize during exercise.
Safety and tolerability assessed by nature, frequency, and severity of Adverse Events (AEs) | Baseline up to week 7
  Adverse Events (AEs) will be coded using medical dictionary for regulatory activities (MedDRA). An AE is any untoward medical occurrence in a participant, temporally associated with the use of investigational product (IP), whether or not considered related to the IP. An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease (new or exacerbated) temporally associated with the use of IP. This includes events related to the comparator and events related to the (study) procedures.
Number of Participants With Laboratory Value Abnormalities and/or Adverse Events (AEs) | Baseline up to week 7
  Number of participants with potentially clinically significant laboratory values.
Number of Participants With Vital Sign Abnormalities and/or Adverse Events (AEs) | Baseline up to week 7
  Number of participants with potentially clinically significant vital signs values.
Number of Participants With 12-lead Electrocardiogram (ECG) Abnormalities and/or Adverse Events (AEs) | Baseline up to week 7
  Number of participants with potentially clinically significant 12-ECG values.
Number of participants with suicidal ideation and/or behavior as assessed by Columbia-Suicide Severity Rating Scale (C-SSRS) | Baseline up to week 7
  The Columbia-Suicide Severity Rating Scale (C-SSRS) is a clinician administered assessment tool that evaluates suicidal ideation and behavior. Number of participants that have an affirmative response provided to the 5 items for suicidal ideation (1. Wish to be dead, 2. Non-specific active suicidal thoughts, 3. Active suicidal ideation with any methods (not plan) without intent to act, 4. Active suicidal ideation with some intent to act, without specific plan, 5. Active suicidal ideation with specific plan and intent) and/or to the 6 items for suicidal behavior (1. Actual attempt, 2. Interrupted attempt, 3. Aborted attempt, 4. Preparatory acts or behavior, 5. Suicidal Behavior 6. Completed suicide,) will be reported.

SECONDARY OUTCOMES:
Change from baseline in systemic oxygen extraction (SOE) | Baseline and Week 6
  Systemic oxygen extraction is defined as the difference between the arterial and venous concentrations of oxygen.
Change from baseline in percent predicted VO2max during aCPET | Baseline and Week 6
  Predicted V02max is measured by the maximum oxygen uptake at peak exercise.
Change from baseline in workload at peak during aCPET | Baseline and Week 6
  Change from baseline in workload at peak during aCPET
Change from baseline in workload at ventilatory anaerobic threshold (VAT) during aCPET | Baseline and Week 6
  Change from baseline in workload at ventilatory anaerobic threshold (VAT) during aCPET
Change from baseline in multivariable gas exchange index (MGI) during SHAPE Test. | Baseline and Week 6
  Change from baseline in multivariable gas exchange index (MGI) during SHAPE Test. The SHAPE Test is a noninvasive exercise test of the functional status of participants.

CONTACTS AND LOCATIONS:
Overall Officials: Senior Medical Director, Study Director — Astellas Pharma Global Development, Inc.
Locations (1):
- Brigham and Women's Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No
Access to anonymized individual participant level data will not be provided for this trial. Further details on Astellas' data sharing policy can be found at https://www.clinicaltrials.astellas.com/transparency/.

REFERENCES:
- See also: Link to plain language summary of the study on the Trial Results Summaries website — https://www.trialsummaries.com/Study/StudyDetails?id=14612&tenant=MT_AST_9011